CLINICAL TRIAL: NCT01010269
Title: A Prospective Controlled Multi-center Study on Vanguard Complete Knee and Vanguard High Flex RP Knee
Brief Title: Vanguard Complete Knee Versus Vanguard High Flex Rotating Platform (RP) Knee Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT.CR.RROW1
Record Dates: First submitted 2009-10-26; First posted 2009-11-10 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanguard Complete Knee (Active Comparator): Vanguard Completed Knee with Microplasty Tibial Tray is designed to hold the tibial knee bearings in a microplsty knee procedure. The Co-Cro-Mo trays are designed with a shorter stem.
  Interventions: Device: Vanguard Complete Knee
- Vanguard High Flex RP (Active Comparator): VGRD High Flex RP knee is an extension to the exsting Vanguard Knee and has been specifically desinged to facilitate greather than 135 degrees of knee flextion as required by certain patients.
  Interventions: Device: Vanguard High Flex RP

INTERVENTIONS:
Device: Vanguard Complete Knee — Vanguard Knee is a metal and polyethylene system indicated for cemented tibial and femoral use.
  Arms: Vanguard Complete Knee
Device: Vanguard High Flex RP — Vanguard High Flex RP is an extension to the existing Vanguard Knee and has been specifically designed to facilitate greater than 135 degrees of knee flexion.
  Arms: Vanguard High Flex RP

SUMMARY:
The purpose of this study is to compare Vanguard High Flex Rotating Platform to Vanguard Complete Knee System in Asian population in terms of early range of motion (ROM), clinical outcomes, and kinetic and kinematic characteristics in relation to healthy knees.

DETAILED DESCRIPTION:
The primary objectives of this clinical study include:

* Evaluate size fit and long term performance of Vanguard Complete Knee ("Fixed") System in Asian and Latino population in comparison to competitor's similar product.
* Evaluate efficacy of Vanguard Complete Knee with Microplasty Tibial Tray.
* Compare Vanguard High Flex Rotating Platform ("High Flex") Knee System to Vanguard Complete Knee System in Asian population in terms of:

  * Early ROM
  * Clinical outcomes
  * Kinetic and Kinematic characteristics in relation to Healthy Knees. o
* Compare current design to new design of Vanguard High Flex Rotating Platform Knee System in terms of :

  * Early ROM
  * Clinical outcomes
  * Kinetic and Kinematic characteristics

ELIGIBILITY:
Inclusion Criteria:

* Painful and disabled knee joint resulting form osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, or arthrodesis.
* Need to obtain pain relief and improve function.
* Ability and willingness of the patient to follow instructions, including control of weight and activity level.
* Good nutritional state of the patient.
* Patient must have reached full skeletal maturity.

Exclusion Criteria:

* Infection, sepsis, osteomyelitis, and failure of previous joint replacement.
* Uncooperative patient or patients with neurologic disorders who are incapable of following directions.
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
American Knee Society Knee Score | 1 Year postop
  Including ROM

SECONDARY OUTCOMES:
Kinematic Fluoroscopic Analysis | 3 yr
  Kinematic Fluoroscopic Analysis
Gait Lab Analysis | 3 yr
  Gait Lab Analysis
EQ5D | 3 mo, 6 mo, 1 yr, 3 yr, 5 yr, 7 yr, 10 yr
  Quality of Life
Radiographic Assessment | immediate postop, 3 mo, 6 mo, 1 yr, 3 yr, 5 yr, 7 yr, 10 yr
  Radiographic Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Chul Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Chul-Won Ha, M.D., Ph.D., Principal Investigator — Samsung Medical Center; Seong-Il Bin, M.D., Ph.D., Principal Investigator — Asan Medical Center; Yong In, M.D., Ph.D., Principal Investigator — Catholic University Uijungbu St. Mary's Hospital
Locations (4):
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Nat'l Uni. Hospital, Seoul
  - The Catholic Uni. of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT01010269/Prot_SAP_000.pdf